CLINICAL TRIAL: NCT05325099
Title: Study of the Effect of Demethylating Agent Azacitidine on Prevention of Acute Kidney Injury-chronic Kidney Disease Continuum
Brief Title: Demethylating Agent Azacitidine on Prevention of Acute Kidney Injury-chronic Kidney Disease Continuum
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202110100MINA
Record Dates: First submitted 2022-04-05; First posted 2022-04-13 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Acute Kidney Disease
MeSH Terms: interventions — Azacitidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AKI patient with azacitidine treatment (Experimental): azacitidine (subcutaneous injection)
  Interventions: Drug: Azacitidine
- AKI patient with placebo treatment (Placebo Comparator): Placebo drug (subcutaneous injection)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azacitidine — azacitidine (Vidaza) 1mg/BW(kg) (subcutaneous injection) QOD x 3 times
  Other Names: Vidaza
  Arms: AKI patient with azacitidine treatment
Drug: Placebo — Placebo (subcutaneous injection) QOD x 3 times
  Arms: AKI patient with placebo treatment

SUMMARY:
Acute kidney injury (AKI) is increasing worldwide in recent years and is a major risk factor of chronic kidney disease (CKD). AKI, acute kidney disease (AKD) and CKD form a continuum whereby initial kidney injury leads to ongoing renal injury and eventually end-stage renal disease if no effective treatment is applied. Nevertheless, there are no useful pharmacotherapies approved clinically for the treatment of AKI and subsequent CKD.

Previous studies of the investigators have confirmed that pericytes are the primary cell source of scar-producing myofibroblasts. Furthermore, the investigators had demonstrated that significant epigenetic modification in transcriptome analysis of pericytes develops in different stage of AKI-CKD continuum. These epigenetic memory made pericytes obtain proliferative and pro-fibrotic phenotypes in activated status and persist in inactivated status. Demethylation by azacitidine prevented AKI-CKD transition, and attenuated fibrogenesis induced by a second adenine-AKI.

Azacitidine has been approved in the United States Food and Drug Administration and European Union for treatment of adult acute myeloid leukemia (AML), particularly recommended front-line treatment for older patients with acute myeloid leukemia who are not candidates for intensive treatment regimens. Dosage of azacitidine in clinical trial is calculated according to previous study and is lower than chemotherapeutic dose. Low dose azacitidine has demethylation effect and less cytotoxicity.

CSA-AKI is the second commonest cause of AKI in ICU. The investigators plan to initiate a double-blind randomized controlled trial (RCT) to recruit CSA-AKI patients. The patients will be divided as azacitidine group and placebo group. Patients in azacitidine group will receive three doses of low dose azacitidine in one week when AKI is diagnosed. After that, the investigators will follow up their renal function and urine protein every three month. Primary composite outcomes include a decline of at least 50% in the estimated GFR, an increase of urine protein-creatinine ratio (UPCR) over 1000 mg/g, and the development of end stage renal disease (ESRD). Secondary outcome is overall mortality.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is increasing worldwide in recent years and is a major risk factor of chronic kidney disease (CKD). An episode of AKI is not only associated with significant risk of short- and long-term morbidity and mortality but also a tremendous burden to patients, societies, and health care system. AKI, acute kidney disease (AKD) and CKD form a continuum whereby initial kidney injury leads to ongoing renal injury and eventually end-stage renal disease if no effective treatment is applied. Nevertheless, there are no useful pharmacotherapies approved clinically for the treatment of AKI and subsequent CKD. Current management can only focus on avoiding risk factors to prevent AKI and supportive care after diagnosis of AKI.

Pericytes, sharing developmental origins with fibroblasts, are the collagen-producing cells contacted with the microvascular. Previous studies of the investigators have confirmed that pericytes are the primary cell source of scar-producing myofibroblasts. Furthermore, the investigators had demonstrated that significant epigenetic modification in transcriptome analysis of pericytes develops in different stage of AKI-CKD continuum. These epigenetic memory made pericytes obtain proliferative and pro-fibrotic phenotypes in activated status and persist in inactivated status. The investigators found methylation of Ybx2 gene and other four repressor genes of αSMA were induced by TGF-b1 after AKI. Demethylation by azacitidine recovered the microvascular stabilizing function of aPericytes, reversed the profibrotic property of iPericytes, prevented AKI-CKD transition, and attenuated fibrogenesis induced by a second adenine-AKI. As a result, azacitidine is a potential therapeutic agents to prevent AKI-CKD continuum by its demethylating effect.

Azacitidine has been approved in the United States Food and Drug Administration and European Union for treatment of adult acute myeloid leukemia (AML), particularly recommended front-line treatment for older patients with acute myeloid leukemia who are not candidates for intensive treatment regimens. Azacitidine is used in clinical trial of other malignancies such as breast cancer or lung cancer. Dosage of azacitidine is calculated according to previous study and is lower than chemotherapeutic dose. Low dose azacitidine has demethylation effect and less cytotoxicity.

CSA-AKI is the second commonest cause of AKI in ICU. 8.2% patients after cardiac surgery in our hospital had severe AKI defined as Kidney Disease Improving Global Outcomes (KDIGO) criteria stage 2 or 3. Therefore, the investigators plan to initiate a double-blind randomized controlled trial (RCT) to recruit CSA-AKI patients. The patients will be divided as azacitidine group and placebo group. Patients in azacitidine group will receive three doses of low dose azacitidine in one week when AKI is diagnosed. After that, the investigators will follow up their renal function and urine protein every three month. Primary composite outcomes include a decline of at least 50% in the estimated GFR, an increase of urine protein-creatinine ratio (UPCR) over 1000 mg/g, and the development of end stage renal disease (ESRD). Secondary outcome is overall mortality. If the results demonstrated the benefit of azacitidine on the prevention of AKI-CKD continuum, the investigators can optimize the strategies and guideline of post-AKI care and the incidence of CKD and ESRD will decrease.

ELIGIBILITY:
Inclusion Criteria:

* Patient with cardiac surgery associated-AKI, stage 2 and stage 3

Exclusion Criteria:

* Chronic kidney disease
* Decompensated heart failure (EF < 45%)
* Liver cirrhosis, child B or C
* Acute infection
* Acute bleeding
* Long-term use of immunosuppressant other than azacitidine
* Patients with active cancer other than acute leukemia or myelodysplastic syndrome
* Leukopenia, anemia or thrombocytopenia
* Pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Renal composite outcome | 2 years after recruitment
  1. A decline of at least 50% in the estimated GFR (compared with baseline eGFR)
  2. An increase of UPCR over 1000 mg/g
  3. The onset of end-stage kidney disease

SECONDARY OUTCOMES:
Overall mortality and cardiovascular death | 2 years after recruitment

CONTACTS AND LOCATIONS:
Overall Officials: Yu Hsiang Chou, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Yu Hsiang Chou, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No